CLINICAL TRIAL: NCT06501976
Title: An Exploratory Study of Lurbinectedin With Radiotherapy in Locally-advanced SCLC After First-line Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4493
Record Dates: First submitted 2024-06-29; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Treatment: Lurbinectedin combined with Thoracic Radiotherapy (Experimental): Patients receive 2 cycles of lurbinectedin 2.6 mg/m2 combined with thoracic radiotherapy followed by 2 cycles of lurbinectedin 2.6 mg/m2 alone. Patients receive lurbinectedin intravenously (IV) over 1 hour on day 1 of each cycle.
  Interventions: Drug: Lurbinectedin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Lurbinectedin — 2.6 mg/m2 , Given IV, every 21 days
  Other Names: PM01183; Zepzelca
Radiation: Radiation Therapy — Thoracic radiotherapy

SUMMARY:
This exploratory trial aims to determine if it is safe to use radiotherapy and lurbinectedin to treat locally-advanced SCLC after first-line therapy. This study will enroll patients with thoracic disease but no distant metastases after first line treatment failure. Lurbinectedin kills tumor cells by blocks transcription and damages the deoxyribonucleic acid (DNA) of tumor cells, which is similar to the way radiation kills tumor cells. Traditional chemotherapy and radiotherapy is a routine medical treatment for locally-advanced SCLC, but the combination is always toxic. This trial may help understand if treating patients with lurbinectedin and radiotherapy could cause less side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To describe the safety in terms of radiation therapy (RT) in combination with lurbinectedin in patients with locally-advanced SCLC after first-line therapy.

SECONDARY OBJECTIVES:

To evaluate the preliminary efficacy of RT plus lurbinectedin, as assessed by Progression free survival (PFS) and Overall survival (OS).

OUTLINE:

Patients receive 2 cycles of lurbinectedin combined with thoracic radiotherapy followed by 2 cycles of lurbinectedin alone. Patients receive lurbinectedin intravenously (IV) over 1 hour on day 1 of each cycle. G-CSF（Granulocyte Colony-Stimulating Factor） will be used for prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Has fully understood this study, voluntarily signed a written informed consent form, and is able to comply with the requirements and restrictions listed in the informed consent form;
* Age ≥ 18 years, Male/female participants;
* Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2;
* With pathologically confirmed diagnosis of Limited Stage SCLC(LS-SCLC),with local progression (mainly thoracic progression) after first-line chemotherapy with or without immunotherapy, but without distant metastasis; (Currently immunotherapy + chemotherapy is not the standard treatment for LS-SCLC);
* Has sufficient bone marrow, liver, kidney, and metabolic function, i.e., the functional levels of organs meet the following requirements:
* Platelets (PLT) ≥ 100×10^9/L;
* Hemoglobin (Hb) ≥ 90 g/L;
* Absolute neutrophil (ANC) ≥ 2.0×10^9/L;
* Regardless of whether liver metastasis is present, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0× upper limit of normal (ULN);
* Alkaline phosphatase (ALP) ≤ 5×ULN;
* Total bilirubin (TBIL) ≤ 1.5×ULN, and direct bilirubin ≤ 1.0×ULN;
* Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 30 mL/min (calculated using the Cockcroft-Gault formula);
* Creatine phosphokinase (CPK) ≤ 2.5×ULN;
* Albumin ≥ 3.0 g/dL.
* A female of childbearing potential (FCBP) must have a negative serum pregnancy test prior to study entry. Woman of childbearing potential (WOCBP) must use adequate contraception during the test drug treatment period and for 6 months after the final dose. Male patients (with partners of WOCBP) must use adequate contraception for the duration of study participation, and 4 months after completion of administration.

Exclusion Criteria:

* With concurrent brain metastasis, a history of spinal cord compression, or meningeal metastasis;
* With bone metastases;
* Patients with obstructive atelectasis, superior vena cava syndrome requiring surgical/ endoscopic/ interventional treatment; suspected or confirmed pulmonary embolism patients; those with uncontrollable large amounts of pleural effusion, ascites, or pericardial effusion;
* Patients known to be allergic to any component of the test drug;
* Pregnancy or breastfeeding or WOCBP who has a positive serum pregnancy test;
* Comorbidities Requirements:

  1. Has unstable angina, myocardial infarction, congestive heart failure (CHF) classified as New York Heart Association (NYHA) II or higher, or other clinically significant cardiovascular diseases currently or within the past year prior to screening;
  2. Patients with uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), or a history of hypertensive crisis or hypertensive encephalopathy;
  3. Patients with severe arrhythmias requiring medication;
  4. Patients with active infections requiring systemic antibacterial, antifungal, or antiviral treatment within 2 weeks prior to administration;
  5. Patients with evidence of bleeding tendencies or coagulation disorders;
  6. Patients with other significant diseases judged unsuitable for entry by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events of radio therapy with lurbinectedin | 30 days following treatment completion
  ≥grade 4 treatment related adverse events within 30 days of final RT fraction; Any treatment related adverse events leading to dose delays or reductions of lurbinectedin; Any treatment related serious adverse events .

SECONDARY OUTCOMES:
Progression free survival (PFS) | From protocol treatment initiation to disease progression or death, assessed up to 24 months
  PFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median PFS will be estimated.
Overall survival (OS) | From treatment initiation to death, , assessed up to 24 months
  OS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median OS will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared